CLINICAL TRIAL: NCT04942301
Title: PhaseⅠStudy to Evaluate PK, Safety, and Preliminary Efficacy of Endostar Standard-dose Intravenous Infusion and Continuous (Pump) Infusion in Combination With 1st-line Platinum-based Doublet Chemotherapy in Patients With Advanced NSCLC
Brief Title: PK Study for Endostar Continuous Intravenous Infusion in NSCLC Patients With 1st-line Platinum Based Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIM-1904-04-ENDO-101
Record Dates: First submitted 2021-05-31; First posted 2021-06-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Endostatins; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endostar pump for three days (Experimental): Group A: The first cycle, Endostar 7.5mg/m2/day, intravenous infusion for 4 hours, D1-14 First 2-4 cycles, Endo 105mg/m2/cycle D1 starts intravenous pump for 72 hours;
  Interventions: Drug: Endostar; Device: use the vein pump to pump drugs; Combination Product: combination therapy
- Endostar pump for seven days (Experimental): Group B: Cycle 1, Endo 7.5mg/m2/day, intravenous infusion for 4 hours, D1-14 First 2-4 cycles, Endo 105mg/m2/cycle D1 starts intravenous pump injection for 168 hours;
  Interventions: Drug: Endostar; Device: use the vein pump to pump drugs; Combination Product: combination therapy

INTERVENTIONS:
Drug: Endostar — This product combined with other combined chemotherapeutics is used to treat patients with stage III/IV NSCLC who are newly treated or relapsed
  Other Names: recombinant human endostatin injection
Device: use the vein pump to pump drugs — During the first 14 days of the first cycle, the experimental drug was pumped daily with an intravenous pump. During cycles 2-4, subjects in group A were pumped with experimental drugs for 3 days and subjects in group B were pumped with experimental drugs for 7 days.
  Other Names: vein pump
Combination Product: combination therapy — Combination therapy with chemotherapy drugs was used

SUMMARY:
This trial is an open-label, randomized, multicenter study to explore Endostar in combination with standard platinum-based chemotherapy with different methods in patients with advanced/metastatic non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
Patients in group A received a standard 21-day treatment cycle of platinum-containing two-drug chemotherapy and endurance treatment. Yep The first cycle of the degree of use is 7.5mg/m2/day intravenous infusion for 4 hours (referred to as the time window of 4h 20min From the 1st day to the 14th day (D1-14 Endo cycle 2-4 uses 105mg/m2/cycle From the first day, continuous intravenous pump injection for 72 hours (the set time window is 72h±2h.).

Patients in group B received a standard 21-day treatment cycle of platinum-containing two-drug chemotherapy and endurance treatment. Yep The first cycle of the degree of use is 7.5mg/m2/day intravenous infusion for 4 hours (referred to as the time window is 4h±20min From the 1st day to the 14th day (D1-14 Endo cycle 2-4 is used 105mg/m2/cycle From the first day, continuous intravenous pump injection for 168 hours (set time window is 168h±2h).

Endostar and chemotherapy drugs are used for 4 cycles. Research will Use RECIST 1.1 standard to evaluate in progress and after enrollment Efficacy assessment will be conducted every 6±1 weeks until the disease progresses, new anti-tumor therapy is started, and the study is withdrawn or At the end of the study, the serum of Endo will be collected in different expected ways to evaluate the pharmacokinetic characteristics; Adverse events were evaluated according to CTCAE5.0 standards. The start time of the test is The first fine was when the informed consent form was signed. The end of the test is the last The subject completed 24 weeks after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in clinical trials and sign an informed consent form.
* Age ≥ 18 years old, including gender.
* Advanced or metastatic NSCLC confirmed by histology and/or cytology: Have not received Systemic chemotherapy for advanced disease (Patients with sensitive mutations such as EGFR and ALK have received corresponding standard alternative treatments, But patients who have not received chemotherapy can be included in the group; have received single-agent PD-L 1 and other immune checkpoint inhibitors Patients, but patients who have not received chemotherapy can enter the group).
* At least one measurable lesion (based on RECIST 1.1).
* ECOG scores 0~1.
* Expected survival time ≥ 3 months.
* The functions of major organs are basically normal, and the laboratory test values during the screening period meet the following standards:

System Laboratory Inspection Standard hematology Absolute neutrophil count >1.5 ×109/L Platelet >100×109/L Hemoglobin >90g/L kidney Serum creatinine or Creatinine clearance rate (CrCl) or glomerular filtration rate (GFR) (Cockcroft-Gault formula) <1.5 × ULN or >60 mL/min1.73m2 (for patients with creatinine level ≥ 1.5 × ULN) liver Total bilirubin (serum) <2.5 × ULN or Direct bilirubin <ULN (for patients with total bilirubin level ≥ 1.5×ULN) AST and ALT <2.5 × ULN or ≤5 × ULN (for patients with liver metastases) Blood clotting International normalized ratio (INR) or prothrombin time (PT) <1.5 × ULN, unless the patient is receiving anticoagulation therapy

Urine routine Urine protein ≤+ (For patients with urine protein ≥++, 24-hour urine protein quantification is required, and 24-hour urine protein needs to be less than 1g)

· Women of childbearing age during the screening period had negative blood pregnancy test results. The patient agrees to self-sign and know Consent to use reliable contraceptive methods within 90 days after the end of treatment.

Exclusion Criteria:

* Patients with uncontrolled primary central nervous system tumors, brain metastases, or meningeal metastases. Patients who were asymptomatic or had their symptoms under treatment (stable and asymptomatic at least 4 weeks after treatment) were allowed to join the group.
* Imaging (CT, PET-CT, or MRI) shows tumors invading large blood vessels.
* It is first clear that pulmonary hemorrhage/hemoptysis (> 1/2 teaspoon about 2.5ml bright red blood) or other clinically significant bleeding symptoms or obvious bleeding possibility occurred in the first 3 months.
* Severe uncontrollable hypertension (defined as systolic blood pressure> 150mmHg and/or diastolic blood pressure> 100mg, or accompanied by hypertensive crisis, hypertensive encephalopathy).
* The QTcF interval of ECG> 480ms within 6 months before the first first time.
* Severe infections within 4 weeks before the first administration require intravenous antibiotics or hospitalization.
* Before the first dose, the adverse events caused by any intervention have not recovered to normal or ≤1 grade. Patients with alopecia (any grade) and sensory neuropathy (≤2 grade) at both ends can be included in the group.
* Received other major surgery besides diagnosis or biopsy within 4 weeks before the first definition.
* 4 weeks or 5 half-lives before the first time (for investigational drugs with known half-lives) internally as a patient Received experimental drug treatment.
* Previously received anti-angiogenic drug treatment.
* Received systemic anti-tumor therapy within 4 weeks before the first dose, including chemotherapy, macromolecular targeting, immunotherapy, and endocrine therapy; within 2 weeks before the first dose or within 5 half-lives of the drug (whichever is longer) ) Receiving small-molecule targeted drug therapy; receiving Chinese/herbal medicine with anti-tumor indications within 2 weeks before the first dose.
* Patients who have received adjuvant chemotherapy within 6 months before the first dose and the disease recurs within 6 months after the start of adjuvant therapy.
* Obvious gastrointestinal bleeding (such as esophageal or gastric varices) or a clear bleeding tendency occurred within 4 weeks before the first dose.
* Those who are allergic to any active or inactive ingredients of Endo or the combined chemotherapeutics.
* Known acute or active hepatitis B, or chronic hepatitis C, or syphilis infection, or human immunodeficiency virus (HIV) infection.
* Patients during pregnancy or lactation.
* Take CYP2C8 substrates (such as repaglinide, rosiglitazone), CYP2C8 inhibitors (such as gemfibrozil), CYP2C8 inducers (such as rifampicin) within 14 days before using the test drug in the first cycle, CYP3A4 substrates (such as midazolam, buspirone, felodipine, lovastatin, eletriptan, sildenafil, simvastatin, triazolam), CYP3A4 inhibitors (such as a Zanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin), CYP3A4 inducer (Such as rifampicin, carbamazepine);
* The researcher believes that the patient has any clinical or laboratory abnormalities or other reasons that are not suitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2021-12-25 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
peak time (Tmax) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
peak concentration (Cmax) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
area under curve (AUC, Including AUC0-t, AUC0-∞) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
terminal elimination half-life (T1/2) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
steady-state minimum blood concentration (CSS min) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
mean steady-state blood concentration (CSS AV) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
accumulation coefficient (RAC) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
mean residence time (MRT) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
apparent volume of distribution (VD) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters
clearance rate (CL) | At the end of the second cycle, each cycle is 21 days
  pharmacokinetic parameters

SECONDARY OUTCOMES:
Adverse events (AE) incidence | through study completion, an average of 1 year
  Adverse event (AE) incidence

OTHER OUTCOMES:
The objective response rate (ORR) | through study completion, an average of 1 year
  The investigator evaluated the objective response rate (ORR), based on the RECIST 1.1 standard
disease control rate (DCR) | through study completion, an average of 1 year
  The investigator evaluated the disease control rate (DCR), based on the RECIST 1.1 standard
the progression-free survival | through study completion, an average of 1 year
  The investigator evaluated the progression-free survival based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Overall Officials: xiaojian zhang, Principal Investigator — the director of the IRB
Locations (1):
- Lan Mu, Shanghai, Shanghai Municipality, China